CLINICAL TRIAL: NCT03223831
Title: Partially Covered Versus Uncovered Pyloro-duodenal Stents for Unresectable Malignant Gastric Outlet Obstruction. A Double Blinded Randomised Controlled Trial.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: National University Hospital, Singapore (Other); Singapore General Hospital (Other); Changi General Hospital (Other); Baldota Institute of Digestive Diseases, Mumbai, India. (Unknown)
Responsible Party: Principal Investigator, Anthony Teoh, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE2016.701-T
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Unresectable Malignant Gastric Outlet Obstruction
Keywords: unresectable malignant gastric outlet obstruction; Partially covered pyloro-duodenal stents; uncovered pyloro-duodenal stents

STUDY DESIGN:
Intervention Model Description: Recruited patients would be randomized to receive either uncovered duodenal stents or partially covered duodenal stents.
Who Masked: Participant
Masking Description: Recruited patients would not be informed of the type of stent that was inserted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially covered duodenal stent (PCDS) (Active Comparator): The PCDS used in the current study is a partially covered metallic pyloro-duodenal stent. It consists of two portions. The stent is 2cm in diameter and the proximal 2cm of the stent is uncovered and flared. The remaining of the stent is covered, where a polytetrafluoroethylene (PTFE) membrane is held between two nitinol mesh.
  Interventions: Other: Partially covered pyloro-duodenal stent
- Uncovered duodenal stent (UDS) (Active Comparator): The UCDS used in the current study is an uncovered stent made of nitinol wire, with a diameter of 20mm. This stent is an unfixed-cell braided stent with low axial force, high flexibility and good conformability.
  Interventions: Other: Uncovered pyloro-duodenal stents

INTERVENTIONS:
Other: Partially covered pyloro-duodenal stent — The PCDS (Niti-S COMVITM - Flare, Taewoong, Gyeonggi-do, South Korea) used in the current study is a partially covered metallic pyloro-duodenal stent. It consists of two portions (Figure 1). The stent is 2cm in diameter and the proximal 2cm of the stent is uncovered and flared. This is designed to provide anchorage of the stent to surrounding tissue and reduce the risk of migration. The remaining of the stent is covered, where a polytetrafluoroethylene (PTFE) membrane is held between two nitinol mesh to prevent the risk of tumour ingrowth into the stent. The stents come in lengths of 6, 8, 10 & 12cm.
  Other Names: PCDS
  Arms: Partially covered duodenal stent (PCDS)
Other: Uncovered pyloro-duodenal stents — The UCDS (Niti-S pyloric-duodenal D stent, Taewoong, Gyeonggi-do, South Korea) used in the current study is an uncovered stent made of nitinol wire, with a diameter of 20mm and length of 6,8,10,12cm. This stent is an unfixed-cell braided stent with low axial force, high flexibility and good conformability.
  Other Names: UCDS
  Arms: Uncovered duodenal stent (UDS)

SUMMARY:
To compare the efficacy of a novel partially covered (PC) versus uncovered (UC) pyloro-duodenal stents (DS) in unresectable malignant gastric outlet obstruction. We hypothesize that the use of PCDS could reduce the re-intervention rates when compared to UCDS.

DETAILED DESCRIPTION:
This would be a prospective multi-centred double-blinded randomised controlled study including all patients suffering from malignant gastric outlet obstruction due unresectable primary gastro-duodenal or pancreatico-biliary malignancies. Five international institutions in Hong Kong, Singapore and India would participate in the study.

The procedure would be performed under conscious sedation or monitored anaesthesia. The patients would be randomised PCDS or UCDS after cannulation of the obstruction site is achieved with the guide-wire. The patients or assessors would be blinded to the type of stent that is inserted.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients ≥ 18 years old
* Confirmed unresectable gastro-duodenal or pancreatico-biliary malignancies
* Suffering from gastric outlet obstruction with a gastric outlet obstruction score of ≤ 1 (appendix 1) 19
* Performance status ECOG ≤3 (appendix 2)

Exclusion Criteria:

* Prior metallic stent placement
* Severe comorbidities precluding the endoscopic procedure (such as cardiopulmonary disease, sepsis, or a bleeding disorder)
* Life expectancy of less than 1 month
* History of gastric surgery
* Linitus plastica
* Coagulation disorders
* Pregnancy
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Re-intervention rate | 1 year
  Percentage of patients requiring additional endoscopic intervention due to stent dysfunction

SECONDARY OUTCOMES:
Technical success | 1 day
  Successful placement of the DS across the site of obstruction, as confirmed by endoscopy or flouroscopy.
Clinical success | 3 days
  Improvement of at least 1 point in the GOOS within 3 days after stent insertion
Adverse events rate | 1 year
  Graded according to the lexicon of endoscopic adverse events
Mortality | 30 days
  Death from any cause
Gastric outlet obstruction scores (GOOS) | 1 year
  Scoring system for food intake
Stent dysfunction | 1 year
  Restenosis of the stent due to tumour ingrowth or overgrowth, stent migration, or fracture
Duration of stent patency | 1 year
  calculated from the time of stent placement to the time of stent dysfunction
Quality of life assessment scores | 1 year
  EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Teoh, FRCSEd(Gen, Principal Investigator — anthoyteoh@surgery.cuhk.edu.hk
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China